CLINICAL TRIAL: NCT03243786
Title: Stay on Track: A Pilot Study of the Effects of Exercise on Mitigating Side Effects and Altering Inflammatory Biomarker Profiles During Radiation Therapy for Breast Cancer
Brief Title: Stay on Track: A Study of Exercise Effects During Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, John Longo, Assistant Professor Radiation Oncology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00027661
Record Dates: First submitted 2017-02-16; First posted 2017-08-09 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week "Stay on Track" intervention (Active Comparator): The study intervention includes three personal exercise training sessions, three dietary counseling sessions, use of a physical activity tracking device, and approximately three weekly text messaging
  Interventions: Behavioral: Lifestyle- Supportive Care
- 12-week self-guided control (Active Comparator): The self guided group does not receive the study intervention, but is offered a Nutrition and wellness guide at the end of 6 months
  Interventions: Behavioral: Lifestyle- Supportive Care

INTERVENTIONS:
Behavioral: Lifestyle- Supportive Care — The intervention examines dietary and activity patterns, body composition, biomarkers and quality of life in breast cancer patients undergoing radiation therapy

SUMMARY:
The purpose of this study is to examine the impact of a lifestyle intervention. The study will examine the Stay on Track program, dietary and activity patterns, body composition, biomarkers and quality of life in breast cancer patients undergoing radiation therapy.

DETAILED DESCRIPTION:
Research Design. The investigators will be conducting an randomized trial in 60 women undergoing radiation treatment for breast cancer to examine the feasibility of a 12-week lifestyle intervention that addresses diet and physical activity and to explore the impact on behavioral, biological and psychosocial outcomes.

Procedure Summary. Patients who are eligible are consented by the research coordinator, after which a baseline assessment will be scheduled. The baseline assessment requires 60 minutes and includes questionnaires, height/weight, dual energy x-ray absorptiometry (DEXA), and phlebotomy. Participants will also wear the Fitbit for one week to establish baseline activity level. After the baseline assessment, women are then randomly assigned to: the 12-week "Stay on Track" lifestyle intervention or the 12-week self-guided control. Both groups complete a post-intervention and a 3-month follow-up visit identical to their baseline assessment. Self-guided controls can utilize their Fitbit and will receive informative binders 24 weeks' post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age;
2. confirmed primary non-metastatic breast adenocarcinoma;
3. planned lumpectomy/segmentectomy/partial mastectomy surgery for primary breast cancer;
4. planning to undergo adjuvant whole breast radiation therapy following a lumpectomy;
5. Have a Karnovsky Performance Score of 70 or above (see Appendix)
6. Patient's Body Mass Index (BMI) is greater than determine by the treating physician, not currently meeting physical activity guidelines: moderate physical activity for at least 30 minutes at least five days a week AND 2 weekly sessions of resistance exercise;
7. have access to a mobile phone with capacity for text messaging (either unlimited or aware and accepting of text messaging charges);
8. understand and speak English;
9. physically able to engage in the intervention;
10. accepting of randomization (Note that anti-estrogen therapy is allowed.)

Exclusion Criteria:

1. Patients who have metastatic disease;
2. Patients with a history of prior malignancy within the past 3 years, other than non-melanoma skin cancer.
3. Patients with serious orthopedic, cardiovascular, or pulmonary conditions, have serious psychiatric or cognitive problems.
4. Patients who have received chemotherapy for their breast cancer.
5. Patients with prior radiotherapy to primary site or adjacent site that results in overlapping radiation fields.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Breast Cancer
Enrollment: 47 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Percent time of personal fitness tracker use during the intervention period for the Stay on Track intervention arm | 6 months

SECONDARY OUTCOMES:
Percent of participant retention thoughout the 12-week intervention through the six month follow-up | 6 months
The percent of eligible patient who choose to take part in the study | 6 months
Number of personal exercise sessions were attended by members in the Stay on Track Intervention Arm | 6 months
Changes in lean soft tissue over the study period associated with intervention and activity | 6 months
Changes in BMI (weight and height will be combined to report BMI in kg/m^2) over the study period associated with intervention and activity | 6 months
Measures of physical activity (self-report and objective) | 6 months
Dietary intake (assessed via Full Length Block Questionnaire) | 6 months
Measures of fatigue (Piper Fatigue Scale Score and physician CTCAE v4.0 Scoring) | 6 months
Measures of skin side effects (CTCAE v4.0 Scoring) | 6 months
Quality of life (FACT-B Questionnaire) over the study period associated with intervention and activity | 6 months
Measures of pain (PROMIS Scale v1.0- Pain Intensity 3a Questionnaire) over the study period associated with intervention and activity | 6 months
Changes in biomarker (GM-CSF) associated with intervention and activity | 6 months
Changes in biomarker (IFN-gamma) associated with intervention and activity | 6 months
Changes in biomarker (IL-1alpha) associated with intervention and activity | 6 months
Changes in biomarker (IL-1beta) associated with intervention and activity | 6 months
Changes in biomarker (IL-4) associated with intervention and activity | 6 months
Changes in biomarker (IL-6) associated with intervention and activity | 6 months
Changes in biomarker (IL-8) associated with intervention and activity | 6 months
Changes in biomarker (IL-10) associated with intervention and activity | 6 months
Changes in biomarker (IL-12) associated with intervention and activity | 6 months
Changes in biomarker (MCP-1) associated with intervention and activity | 6 months
Changes in biomarker (TNF-alpha) associated with intervention and activity | 6 months
Changes in biomarker (adiponectin) associated with intervention and activity | 6 months
Changes in biomarker (leptin) associated with intervention and activity | 6 months
Changes in biomarker (CRP) associated with intervention and activity | 6 months
Changes in blood insulin level associated with intervention and activity | 6 months
Changes in blood hemoglobin A1C level associated with intervention and activity | 6 months
Changes in blood glucose level associated with intervention and activity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Bergom, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No